CLINICAL TRIAL: NCT06945185
Title: Motor Imagery Training for Upper Limb Functional Strength in Chronic Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/64
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Chronic Stroke
Keywords: Motor Imagery; Stroke; Neurorehabilitation; Functional strength
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP A- CONVENTIONAL PHYSICAL THERAPY (Active Comparator): The participants will receive conventional physical therapy focusing on active range of motion, strengthing and coordination exercises.
  Subjects will receive protocol of 45 min thrice a week for 8 weeks with 2 min rest in between.
  The exercises will focus on active range of motion, weight exercises to increase strength and coordination exercises to improve movement coordination.
  Interventions: Procedure: Intervention Group A Conventional Physical Therapy
- INTERVENTION GROUP B- MOTOR IMAGERY WITH CONVENTIONAL PHYSICAL (Experimental): The participants will recieve conventional physical therapy focusing on active range of motion, strengthing and coordination exercises.
  Subjects will recieve protocal of 45 min thrice a week for 8 weeks with 2 min rest in between.
  The exercises will focus on active range of motion, weight exercises to increase strength and coordination exercises to improve movement coordination.
  Interventions: Procedure: Intervention Group B Motor Imagery with Conventional Physical Therapy

INTERVENTIONS:
Procedure: Intervention Group A Conventional Physical Therapy — Active Range of Motion Exercises: (5-10 reps with 2 sets) Finger bends, finger spreads, finger to thumb opposition, thumb to palm stretches, palm up and down, wrist rotation, wrist bends, elbow bends, shoulder shrugging and shoulder rotation.
  Strengthening Exercises: (10-15 reps 2 sets weight 500 ml to 1L water bottle). Finger pinch, power grip, finger spread, pushing movement, wrist curls, roll and squeeze, bicep curls, side arm raise, lifting objects to a height, pulling resistance band.
  Coordination Exercises: (10-15 reps 2 sets) finger to finger, finger to doctor's finger, finger to nose, holding and lifting coins, buttoning, holding and lifting coins, alternate hand movement, closing and opening hand.
  Arms: CONTROL GROUP A- CONVENTIONAL PHYSICAL THERAPY
Procedure: Intervention Group B Motor Imagery with Conventional Physical Therapy — 1. Subjects will be asked to sit comfortably on a chair with a backrest. A Quiet environment is ensured for proper concentration of subject .Take deep breaths for 2-3 min to relax.
  2. Subjects will be asked to close their eyes and imagine the training scene for each task for 5 min while listening to the therapist 's voice describing the motion.
  3. The non-paralysis part of the body's movement was imagined first and then the movement of the paralysis part was imagined.
  4. Upon completion of the mental practice for the first activity, the subject will be given a comfortable break.
  Motor Imagery Training:
  Week 1-2: Approaching and holding a cup, turning book pages and grasping pencil to write.
  Week 3-4: wiping desk, turning door handle and drinking water from cup. Week 5-6: pressing light switch on and off, turning faucet and putting card in wallet.
  Week 7-8: folding towel, brushing teeth and brushing hair. Imagine for 30 sec 2-3 repetitions.
  Arms: INTERVENTION GROUP B- MOTOR IMAGERY WITH CONVENTIONAL PHYSICAL

SUMMARY:
Stroke is a leading cause of upper extremity deficits worldwide. Persistent upper extremity dysfunction affects many post stroke patients and is strongly associated with decreased activities of daily living and poor quality of life.

There is accumulating evidence of a cross-over effect with training of one limb that slightly increase strength and coordination in contralateral untrained limb through neurological adaptations.

One of rehabilitation that is beneficial for stroke patient is motor imagery, a mental rehearsal of a movement that does not include physical movement has been shown to enhance upper limb function.

Evidence demonstrate that MI not only activates motor cortical and subcortical regions but also induces plastic change in motor networks and modulates synaptic activity at spinal level.

DETAILED DESCRIPTION:
OBJECTIVE:

The objectives of this study are:

1. To improve upper limb functional strength.
2. To improve the upper limb coordination.
3. To improve upper limb functional improvement.

HYPOTHESIS

Alternate Hypothesis:

There will be statistically significant difference in effects of motor imagery technique combined with conventional physical therapy and in comparison to conventional physical therapy alone on upper limb functional strength, coordination and functional improvement in chronic stroke. (p<0.05).

Null Hypothesis:

There will be no statistically significant difference in effects of motor imagery technique combined with conventional physical therapy and in comparison to conventional physical therapy alone on upper limb functional strength, coordination and functional improvement in chronic stroke. (p>0.05).

Research Design: Experimental study. Randomized Control Trial

ELIGIBILITY:
Inclusion Criteria:

* Stroke duration 6 months onwards (chronic stroke).
* age 45 years and above.
* Both genders.
* Access cognitive function score > 24 on MoCA.

Exclusion Criteria:

* Patients with any comorbidity, previous surgery and congenital anomly.
* Patient with any fracture/ MSK disorders.
* Score 3 or more on Modified Ashworth scale.
* Patients with hearing impairments

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
FUNCTIONAL STRENGTH | 8 weeks
  FUNCTONAL STRENGTH WILL BE ASSESSED USING WOLF MOTOR FUNCTION TEST
Coordination | 8 weeks
  The Action Research Arm Test (ARAT) will be used to assess upper extremity performance

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan